CLINICAL TRIAL: NCT02348788
Title: Artemether-lumefantrine vs Chloroquine in Patients With Acute Non-severe P. Vivax Malaria in Sabah, Malaysia
Brief Title: Artemether-lumefantrine vs Chloroquine for Uncomplicated P. Vivax Malaria in Malaysia
Acronym: PRIMAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menzies School of Health Research (Other)
Collaborators: Ministry of Health, Malaysia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR91391379918375 ￼
Record Dates: First submitted 2015-01-11; First posted 2015-01-28 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Plasmodium Vivax Malaria Without Complication
Keywords: Vivax; Malaria; artemether-lumefantrine; chloroquine; RCT
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination; Primaquine; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether-lumefantrine + Primaquine (Active Comparator): 1 tablet = 20mg artemether and 120mg lumefantrine. Dosing at 0, 8, 24, 36, 48 and 60 hours. Dose according to bodyweight; >35kg = 2 tablets, 26-35kg = 3 tablets, 16-25kg = 2 tablets, >10-15kg = 1 tablet.
  Primaquine = 7.5mg tablet. Dosing daily for 14 days from Day 0. Dose according to bodyweight; >35kg = 30mg, <35kg = 0.5mg/kg
  Interventions: Drug: Artemether-lumefantrine + Primaquine
- Chloroquine + Primaquine (Active Comparator): 1 tablet contains 155mg chloroquine base. Adult dose (>35kg); 620mg (4 tablets) at 0 hours, and 310mg (2 tablets) at 6-8, 24 and 48 hours.
  Child dose (>10-35kg); 10mg/kg at 0 hours, and 5mg/kg at 6-8, 24 and 48 hours. Primaquine = 7.5mg tablet. Dosing daily for 14 days from Day 0. Dose according to bodyweight; >35kg = 30mg, 10-35kg = 0.5mg/kg
  Interventions: Drug: Chloroquine + Primaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine + Primaquine
  Arms: Artemether-lumefantrine + Primaquine
Drug: Chloroquine + Primaquine
  Arms: Chloroquine + Primaquine

SUMMARY:
Both artemether-lumefantrine and chloroquine are currently used and recommended by Malaysian Ministry of Health as blood stage treatments for non-severe P. vivax and P. knowlesi malaria. Microscopic misdiagnosis between Plasmodium species remains a large issue in Sabah, Malaysia and elsewhere. In order to facilitate potential policy change to a unified ACT guideline for all malaria species in Sabah artemether-lumefantrine needs to be evaluated for P. vivax malaria.

Preliminary data in a recently completed RCT evaluating artesunate-mefloquine vs chloroquine for P. vivax showed up to 36% P. vivax recurrence with chloroquine monotherapy by day 28 post treatment without primaquine. Based on these data blood stage chloroquine treatment failure rates should also be evaluated in the context of standard concurrent (rather than delayed) liver stage primaquine dosing, due to both its potential blood stage synergistic effect in addition to known decreased recurrence rates. As artemether-lumefantrine is one of the current first line Ministry of Health ACTs used in Sabah with a lower adverse event profile compared to artesunate-mefloquine, this was recommended as the more appropriate ACT to evaluate against chloroquine.

DETAILED DESCRIPTION:
Malaria due to infection with P. vivax is currently estimated at up to 390 million episodes per year worldwide, with substantial morbidity caused by the recurrent nature of its infection, associated anaemia and adverse effects on pregnancy, and ability to cause severe disease and death. The majority of malaria cases from all Plasmodium species in Malaysia are from the Eastern state of Sabah, where despite around a 36-fold reduction in incidence since the implementation of malaria eradication programs in 1961, minimum estimates based on unpublished microscopy data from Sabah State public health records still detailed 8685 malaria cases in 2009-2011. While P. vivax accounts for between 30-50% of these figures currently, studies have demonstrated as overall transmission rates in countries previously endemic for malaria decline the proportion of cases attributable to P. vivax increases. Mixed P. falciparum / P. vivax infections are also likely to be underestimated in areas of co-endemicity, with high rates of recurrence of P. vivax shown in studies following treatment for apparent P. falciparum mono-infection or mixed Plasmodium spp. infections.

Malaysian Ministry of Health guidelines currently recommends chloroquine and primaquine as first line treatment for the erythrocytic and hypnozoite life stages of uncomplicated P. vivax malaria respectively. While resistance to chloroquine has previously been documented in Sabah and also Peninsular Malaysia, the unstable transmission dynamics and recent reduction in P. vivax incidence due to public health measures mean the current risk of chloroquine-resistant P.vivax transmission is likely to be low. Despite this, due to documented increasing resistance in surrounding countries including Indonesia, Thailand, Vietnam, and PNG, transient populations of migrant workers, and recent concerns of the failing efficacy of hypnozoite eradication by primaquine, the need for ongoing therapeutic efficacy monitoring is recommended.

There is also growing support for artemisinin-based combination therapy (ACT) as a unified first line treatment choice in areas co-endemic for P. falciparum and P. vivax, as adopted by a small number of countries including PNG, Solomon Islands, Vanuatu and Papua, Indonesia, due to the regional increase of chloroquine-resistant P. vivax, and ongoing concerns over the microscopic misdiagnosis of Plasmodium species. This is also particularly relevant for P. knowlesi malaria, as it is frequently misidentified on microscopy as P. falciparum and P. malariae due to morphological similarities in the early trophozoite, and late trophozoite and schizont life stages respectively, with studies showing up to 80% of P. malariae and 7-12% of P. falciparum in this region are actually P. knowlesi when definitively evaluated with PCR. Misdiagnosis has concerning treatment implications, as although P. knowlesi has been shown to respond well to ACT and chloroquine, unlike P. malariae, knowlesi malaria has a rapid 24-hour replication rate and can cause hyperparasitaemia, severe complications and fatal outcomes, while the inadvertent use of chloroquine for widely chloroquine-resistant P. falciparum may also have fatal consequences.

Previous reluctance to use ACTs in presumed chloroquine-sensitive P.vivax areas were centered on concerns over efficacy and cost. The advent of generically produced ACTs is improving cost-related issues, while a recent Cochrane review of clinical trials looking at the use of ACT versus chloroquine for uncomplicated vivax malaria showed that ACTs are equivalent to chloroquine in preventing recurrent parasitaemia in the first 28 days (RR 1, 95% CI 0.30 to 3.39), and those with long half lives such as mefloquine or piperaquine are superior over a 6-8 week follow up, with fewer recurrent episodes after day 28 (RR 0.47, 95% CI 0.29 to 0.76). This post treatment prophylaxis benefit of longer acting agents extends to the reduction in gametocyte carriage, delay in relapse or re-infection and decreased risk of anaemia development, all of which contribute to decreased transmissibility and health care cost.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 1 year of age and weighing more than 10kg
* Microscopic diagnosis of P. vivax monoinfection
* Negative P. falciparum malaria rapid diagnostic test (histidine-rich-protein 2)
* Fever (temperature ≥37.5°C) or history of fever in the last 48 hours
* Written informed consent to participate in trial

Exclusion Criteria:

* Clinical or laboratory criteria for severe malaria, including warning signs, according to modified WHO 2010 criteria
* Parasitaemia > 100,000 /μL
* Pregnancy or lactation
* Known hypersensitivity or allergy to study drugs
* Serious underlying disease (cardiac, renal or hepatic)
* Received anti-malarials in previous 2 months
* History of psychiatric illness, epilepsy, or cerebral malaria

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Parasite clearance at 48 hours | 48 hours
  The difference in proportion of patients with negative microscopy for P. vivax asexual parasites at 48 hours after treatment with A-L compared to CQ.

SECONDARY OUTCOMES:
Parasite clearance time in hours | Within 72 hours post treatment
  The difference in absolute time in hours post treatment to microscopic parasite clearance between treatment arms
Parasite clearance at day 1 and day 3 | At 24 and 72 hours post treatment
  The difference in proportion of patients with negative microscopy for P. vivax asexual parasites at 24 and 72 hours between treatment arms
Treatment outcome | Day 28 and 42 post treatment
  Early treatment failure (ETF), late treatment failure (LTF), and adequate parasitological and clinical response (APCR) at day 28 and day 42
Risk of anaemia | Day 28 post treatment
  Proportion with haemoglobin less than 12 g/dL in women or less than 13 g/dL in men between treatment arms
Fractional fall in haemoglobin at day 3 | Day 3 post treatment
  Difference in fractional fall in haemoglobin concentration between treatment arms 3 days post treatment
Haemoglobin nadir | 42 days post treatment
  Difference in risk of lowest recorded haemoglobin concentration between treatment arms during 42 day follow-up
Risk of P. vivax gametocyte carriage during follow up | 42 days
  The difference in proportion of microscopic P. vivax gametocyte carriage between treatment arms during 42 day follow up
Risk of adverse events | 42 days
  Risk of adverse events (AE) and serious adverse events (SAE) including relationship to study drugs throughout follow up
Length of hospital inpatient stay | From 2-9 days post enrolment
  Number of days post enrolment requiring admission until treatment completed and 2 negative blood slides for malaria allowing discharge as per Malaysian Ministry of Health guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Timothy William, MBBS, FRCP, Principal Investigator — Ministry of Health, Malaysia
Locations (3):
- Malaysia (3):
  - Kota Marudu District Hospital, Kota Marudu, Sabah
  - Kudat District Hospital, Kudat, Sabah
  - Pitas District Hospital, Pitas, Sabah

IPD SHARING:
Plan to Share IPD: Undecided